CLINICAL TRIAL: NCT01455350
Title: Efficacy of Treatments for Provoked Vestivulodynia : a Randomised Clinical Trial Comparing Multimodal Physiotherapy Treatments to Topical Lidocaine
Brief Title: Efficacy of a Physiotherapy Treatment in Women Suffering From Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Mélanie Morin, Physiotherapist, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOP-115028
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Vestibulodynia
Keywords: provoked vestibulodynia; multimodal physiotherapy; lidocaine
MeSH Terms: conditions — Vulvodynia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): 10 week treatment of daily application of topical lidocaine
  Interventions: Drug: lidocaine
- Multimodal physiotherapy (Experimental): 10 weeks of weekly multimodal physiotherapy treatments
  Interventions: Procedure: Multimodal physiotherapy

INTERVENTIONS:
Procedure: Multimodal physiotherapy — 10 weeks of weekly physiotherapy treatments including relaxation techniques, stretching and pelvic floor muscle control exercises.
  Arms: Multimodal physiotherapy
Drug: lidocaine — 10 weeks of daily topical 5% lidocaine application
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
Chronic gynaecological pain is a major medical problem that affects 20-30% of women at different moments of their life. This largely neglected issue has a significant impact on the sexual and conjugal life of women suffering from it as well as on their psychological health. Furthermore, this kind of pain is not well understood, often misdiagnosed or even totally ignored. Also, treatment is limited and not extensively studied. This study aims at better understanding and treating gynaecological pain. The focus of the study will be provoked vestibulodynia, pain at the entry of the vagina. The efficacy of specialized pelvic floor physiotherapy will be compared to a topical cream (lidocaine) applied to the vulva. The treatment efficacy will be assessed in 234 women (aged from 18-45 years old) suffering from provoked vestibulodynia recruited in 4 hospitals (CHUS, Jewish General Hospital, Royal-Victoria Hospital, CHUM St-Luc).

DETAILED DESCRIPTION:
This is a randomised controlled trial comparing the impact of multimodal physiotherapy treatments to topical lidocaine in women suffering from provoked vestibulodyina. The first treatment consists of 10 sixty minutes weekly physiotherapy treatments including relaxation techniques, stretching and pelvic floor muscle control exercises. The second treatment is a night time application of lidocaine to the vulva for 10 weeks. Physiotherapists will then evaluate women's pain and sexual function right after the treatment and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain in at least 90% of sexual intercourses.
* Moderate to severe pain during the cotton-swab test at one of more vestibule regions (5/10 minimum pain evaluation on the verbal pain intensity scale).
* Pain limited to the vestibule during vaginal penetrations and during activities applying pressure on the vestibule.
* Provoked vestibulodynia lasting at least 6 months prior to the study and diagnosed by a standardised gynaecologic exam protocol by one of our collaborator.

Exclusion Criteria:

* Major psychiatric condition or pelvic pathology associated with a genital pain problem (e.g.: dyspareunia).
* Use of medication that could influence pain perception.
* Actual or past pregnancy.
* Vulvar or vaginal surgery
* Post-menopausal state
* Unwillingness to restrain from other treatments till the 6 months post-treatment evaluation.
* Urogynaecologic symptoms (urinary/anal incontinence, pelvic organs prolapsus, urinary/vaginal infection active or during the last 3 months).
* Incapacity to have sexual intercourse including vaginal penetration during the last 6 months.
* Physiotherapy treatments or lidocaine application prior to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in pain during intercourse | before treatment, after treatment, 6 months after treatment
  evaluated with a visual analog scale
Change in global sexual function | before treatment, after treatment, 6 months after treatment
  evaluated with the female sexual function index (FSFI)

SECONDARY OUTCOMES:
Change in pain catastrophizing | before treatment, after treatment, 6 months after treatment
  evaluated using the pain catastrophizing scale
Change in psychologic distress | before treatment, after treatment, 6 months after treatment
  evaluated using the State-trait Anxiety Inventory (STAI)
Change in fear of pain | before treatment, after treatment, 6 months after treatment
  evaluated using the Pain Anxiety Symptoms Scale (PASS-20)
Change in vulvar blood circulation | before treatment, after treatment, 6 months after treatment
  evaluated using a doppler laser
Change in pelvic floor muscles function | before treatment, after treatment, 6 months after treatment
  evaluated using transperineal ultrasound and dynamometry
Change in pain sensitivity (pressure pain) | before treatment, after treatment, 6 months after treatment
  evaluated using a vulvagesiometer

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Morin, Pht, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - University of Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Background] Morin M, Dumoulin C, Bergeron S, Mayrand MH, Khalife S, Waddell G, Dubois MF; Provoked vestibulodynia (PVD) Study Group. Randomized clinical trial of multimodal physiotherapy treatment compared to overnight lidocaine ointment in women with provoked vestibulodynia: Design and methods. Contemp Clin Trials. 2016 Jan;46:52-59. doi: 10.1016/j.cct.2015.11.013. Epub 2015 Nov 18. PMID 26600287
- [Result] M. Morin, C. Dumoulin, S. Bergeron, M.H. Mayrand, S. Khalifé, G. Waddell, O. Dubois, M.F. Dubois, PVD Study Group. Randomized controlled trial of multimodal physiotherapy treatment compared to overnight topical lidocaine in women suffering from provoked vestibulodynia. 40th Annual Meeting of the International Urogynecological Association, Nice, France, 2015, Int Urogynecol J, 1(Supp - June 2015), PP22.
- [Derived] Morin M, Dumoulin C, Bergeron S, Mayrand MH, Khalife S, Waddell G, Dubois MF; PVD Study Group. Multimodal physical therapy versus topical lidocaine for provoked vestibulodynia: a multicenter, randomized trial. Am J Obstet Gynecol. 2021 Feb;224(2):189.e1-189.e12. doi: 10.1016/j.ajog.2020.08.038. Epub 2020 Aug 18. PMID 32818475
- [Derived] Benoit-Piau J, Dumoulin C, Carroll MS, Mayrand MH, Bergeron S, Khalife S, Waddell G, Morin M; Provoked Vestibulodynia (PVD) Study Group. Efficiency and Cost: E-Recruitment Is a Promising Method in Gynecological Trials. J Sex Med. 2020 Jul;17(7):1304-1311. doi: 10.1016/j.jsxm.2020.04.005. Epub 2020 May 17. PMID 32434709